CLINICAL TRIAL: NCT02442726
Title: Activation of A-delta-fibres and C-fibres in a First Degree Thermal Injury in Volunteers
Acronym: BI-Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, mads u werner, MD, PhD, DMSc, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-2-2014-002
Record Dates: First submitted 2015-05-03; First posted 2015-05-13 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Subjects
Keywords: Heat Injury; Humans; Laser Stimulation; Quantitative Sensory Testing; Reaction Time; Secondary Hyperalgesia; Thermal Thresholds
MeSH Terms: conditions — Hyperalgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thermal Injury (Active Comparator): A first degree heat injury is induced by a contact thermode (12.5 cm2; 47C; 420 s) applied at the skin at the lower leg. CO2-Laser stimulation (Laser Stimulation Device, SIFEC)
  Interventions: Device: CO2-Laser stimulation (Laser Stimulation Device, SIFEC)
- Sham Injury (Sham Comparator): A sham "injury" is induced by a contact thermode (12.5 cm2; 38C; 420 s) applied at the skin at the lower leg. CO2-Laser stimulation (Laser Stimulation Device, SIFEC) is used to assess
  Interventions: Device: CO2-Laser stimulation (Laser Stimulation Device, SIFEC)

INTERVENTIONS:
Device: CO2-Laser stimulation (Laser Stimulation Device, SIFEC) — Laser stimuli are evenly applied in 15 spots (each 6 mm in diameter) in the primary hyperalgesic zone (application zone of the contact thermode) and in the secondary hyperalgesic zone (1 cm outside the application zone of the contact thermode).

SUMMARY:
The aim of this study is to measure reaction times and thermal detection thresholds to CO2 laser stimulation of the skin, before and after a first degree thermal injury, in the primary and secondary hyperalgesia area, in order to investigate whether different nerve-fiber classes are activated in the post-injury phase. The study results are expected to uncover existence of a peripheral inflammatory input contributing to secondary hyperalgesia.

DETAILED DESCRIPTION:
BACKGROUND The conduction speed of peripheral nerve fibers depends on the nerve diameter. The conduction velocity of large myelinated fibers are 50 - 120 m/s, while for the smaller myelinated A-delta- and unmyelinated C-fibers, they are in the range of 5-10 m/s, and 0.5-1 m/s, respectively. Applying short laser pulses with a high energy density and synchronization, simple reaction times can be used to determine the type of fiber class that has been activated. Research from the group of Plaghki and colleagues has shown that when stimulating surface areas are between 15 and 50 sq.mm at a supra-threshold intensity for activating A-delta-fibers, a typical bimodal response pattern is observed with a first peak centered around 400 ms and a second around 850 ms. Whereas the early peak is due to activation of A-delta-fibers, the second peak is caused by C-fiber activation.

HYPOTHESIS Following a mild thermal skin injury (47ºC, 420 s, 9.0 or 12.5 sq.cm area) the injured area is associated with erythema and an increased sensitivity, i.e. pain is easily evoked by mechanical and thermal stimuli in the primary hyperalgesia area. In normal skin surrounding the injury mechanical and thermal allodynia and hyperalgesia, are present. Innocuous stimuli in this secondary hyperalgesia area may elicit pain. This is believed to be a central process suggested by pioneering research in the 1980s and 1990s. The term for this phenomenon is heterosynaptic central facilitation meaning that innocuous stimuli may activate normally high-threshold nociceptive dorsal horn neurons leading to allodynia. This conversion of an innocuous stimulus in normal skin just outside of the injury, to a pain generating stimulus, is the result of a change in the sensory processing within the CNS. This processing is probably regulated by spino-bulbo-spinal loops including the rostral ventro-medial medulla (RVM) and locus coeruleus (LC).

The study hypotheses are, first, that the reaction times at the thermal injury site (i.e. primary hyperalgesia area) are changed compared to the pre-injury level. Second, that the sensory changes in the secondary hyperalgesia area, following a thermal injury, are not exclusively centrally mediated, but that also changes in peripheral afferents, e.g. A-delta-fibers (AMH type I) are demonstrable by assessments of reaction times to CO2 laser pulses.

A well-known alternative to laser stimulation is the use of a contact thermode with a much larger stimulation area, i.e. 2.5 to 16 sq.cm. The substantially larger area of the contact thermode, combined with a slower heating rate, compared to the laser stimulus (< 0.5 sq.cm, 10 ms), may induce pronounced spatial and temporal summation, interfering with accurate interpretation of sensory data. A recent method-comparison study in patients with postherpetic neuralgia, comparing assessments obtained by a contact thermode (9 sq.cm) and by laser stimuli (< 0.25 sq.mm), indicates that the laser method is more sensitive and specific in detecting thermal sensory abnormalities. Since the laser stimulus gives a steeper slope of heating profile and a more synchronized activation of warmth- and heat-sensitive small fibers, i.e. C- and A-delta-fibers, in the skin laser stimulation is the preferred method in the present study.

CLINICAL IMPLICATIONS The propensity for developing secondary hyperalgesia may reflect a predisposition for developing persistent postsurgical pain. It has been estimated that 2-10% of patients undergoing otherwise uncomplicated surgical procedures will suffer from persistent postsurgical pain. Investigating the pathophysiological mechanisms behind secondary hyperalgesia may therefore increase our understanding of the transition to chronic pain and thereby improve our management strategies for this large patient group.

ELIGIBILITY:
Inclusion Criteria:

* healthy right-handed males
* non-smokers (due to fluctuating skin temperatures in smokers)
* normal thermal perception (warmth detection threshold [WDT], cool detection threshold [CDT] and heat pain threshold [HPT])
* familiarized with the thermal injury and quantitative sensory testing
* understands written and verbal study information in Danish
* understands written and verbal study information in English

Exclusion Criteria:

* lesions on the lower leg
* unable to cooperate with the sensory testing
* suspected neurological disease
* hereditary predisposition to peripheral neurological disease
* inability to develop secondary hyperalgesia area (non-responder)14
* "small-area" responder (secondary hyperalgesia area < 36 cm2)
* participated in pharmacological trials during the preceding 4 weeks
* participated in a thermal-injury trial during the preceding 8 weeks
* intake of any medication during the preceding 48 hours
* intake of prescription drugs during the preceding 7 days

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes in distribution of reaction times assessed by laser stimuli in the thermal injury area (the primary hyperalgesia area) comparing post-injury values with pre-injury, baseline values. | 24 hours
  Assessments are performed at Baseline, 1 h post-thermal injury and 24 h post-thermal injury. Changes compared to Baseline are analyzed.
Changes in distribution of reaction times assessed by laser stimuli in the secondary hyperalgesia area comparing post-injury values with pre-injury, baseline values. | 24 hours
  Assessments are performed at Baseline, 1 h post-thermal injury and 24 h post-thermal injury. Changes compared to Baseline are analyzed.

SECONDARY OUTCOMES:
Changes in thermal pain thresholds assessed by laser stimuli in the thermal injury area (the primary hyperalgesia area) comparing post-injury values with pre-injury, baseline values. | 24 hours
  Assessments are performed at Baseline, 1 h post-thermal injury and 24 h post-thermal injury. Changes compared to Baseline are analyzed.
Changes in thermal pain thresholds assessed by laser stimuli in the secondary hyperalgesia area comparing post-injury values with pre-injury, baseline values. | 24 hours
  Assessments are performed at Baseline, 1 h post-thermal injury and 24 h post-thermal injury. Changes compared to Baseline are analyzed.
Thermal detection thresholds assessed by laser stimuli in the thermal injury area (the primary hyperalgesia area) comparing post-injury values with pre-injury, baseline values. | Baseline, 1 h post-thermal injury; 24 h post-thermal injury
Changes in thermal detection thresholds assessed by laser stimuli in the secondary hyperalgesia area comparing post-injury values with pre-injury, baseline values. | 24 hours
  Assessments are performed at Baseline, 1 h post-thermal injury and 24 h post-thermal injury. Changes compared to Baseline are analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Mads U Werner, MD, DMSc, Principal Investigator — Neuroscience Center, Copenhagen University Hospital, Denmark; Ron Kupers, MSc, Study Chair — Panum Institute, Copenhagen University, Denmark; Henrik Kehlet, MD, DMSc, Study Chair — JMC, Copenhagen University Hospital, Denmark
Locations (1):
- BRAINLab, Department of Neuroscience and Pharmacology, Panum Institute, Copenhagen, Denmark

REFERENCES:
- [Background] Pedersen JL, Kehlet H. Hyperalgesia in a human model of acute inflammatory pain: a methodological study. Pain. 1998 Feb;74(2-3):139-51. doi: 10.1016/s0304-3959(97)00160-7. PMID 9520228
- [Background] Naert ALG, Kehlet H, Kupers R. Characterization of a novel model of tonic heat pain stimulation in healthy volunteers. Pain. 2008 Aug 15;138(1):163-171. doi: 10.1016/j.pain.2007.11.018. Epub 2008 Jan 22. PMID 18207325
- [Background] Pedersen JL, Kehlet H. Secondary hyperalgesia to heat stimuli after burn injury in man. Pain. 1998 Jun;76(3):377-384. doi: 10.1016/S0304-3959(98)00070-0. PMID 9718256
- [Background] Torebjork HE, LaMotte RH, Robinson CJ. Peripheral neural correlates of magnitude of cutaneous pain and hyperalgesia: simultaneous recordings in humans of sensory judgments of pain and evoked responses in nociceptors with C-fibers. J Neurophysiol. 1984 Feb;51(2):325-39. doi: 10.1152/jn.1984.51.2.325. PMID 6707724
- [Background] Cook AJ, Woolf CJ, Wall PD. Prolonged C-fibre mediated facilitation of the flexion reflex in the rat is not due to changes in afferent terminal or motoneurone excitability. Neurosci Lett. 1986 Sep 25;70(1):91-6. doi: 10.1016/0304-3940(86)90443-x. PMID 3774223
- [Background] Woolf CJ, Wall PD. Relative effectiveness of C primary afferent fibers of different origins in evoking a prolonged facilitation of the flexor reflex in the rat. J Neurosci. 1986 May;6(5):1433-42. doi: 10.1523/JNEUROSCI.06-05-01433.1986. PMID 3711988
- [Background] Torebjork HE, Lundberg LE, LaMotte RH. Central changes in processing of mechanoreceptive input in capsaicin-induced secondary hyperalgesia in humans. J Physiol. 1992 Mar;448:765-80. doi: 10.1113/jphysiol.1992.sp019069. PMID 1593489
- [Background] LaMotte RH, Lundberg LE, Torebjork HE. Pain, hyperalgesia and activity in nociceptive C units in humans after intradermal injection of capsaicin. J Physiol. 1992 Mar;448:749-64. doi: 10.1113/jphysiol.1992.sp019068. PMID 1593488
- [Background] Werner MU, Petersen KL, Rowbotham MC, Dahl JB. Healthy volunteers can be phenotyped using cutaneous sensitization pain models. PLoS One. 2013 May 9;8(5):e62733. doi: 10.1371/journal.pone.0062733. Print 2013. PMID 23671631
- [Background] Franz M, Spohn D, Ritter A, Rolke R, Miltner WHR, Weiss T. Laser heat stimulation of tiny skin areas adds valuable information to quantitative sensory testing in postherpetic neuralgia. Pain. 2012 Aug;153(8):1687-1694. doi: 10.1016/j.pain.2012.04.029. Epub 2012 May 31. PMID 22657400
- [Background] Arendt-Nielsen L, Chen AC. Lasers and other thermal stimulators for activation of skin nociceptors in humans. Neurophysiol Clin. 2003 Dec;33(6):259-68. doi: 10.1016/j.neucli.2003.10.005. PMID 14678840
- [Background] Martinez V, Ammar SB, Judet T, Bouhassira D, Chauvin M, Fletcher D. Risk factors predictive of chronic postsurgical neuropathic pain: the value of the iliac crest bone harvest model. Pain. 2012 Jul;153(7):1478-1483. doi: 10.1016/j.pain.2012.04.004. Epub 2012 May 2. PMID 22560289
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Johansen A, Schirmer H, Stubhaug A, Nielsen CS. Persistent post-surgical pain and experimental pain sensitivity in the Tromso study: comorbid pain matters. Pain. 2014 Feb;155(2):341-348. doi: 10.1016/j.pain.2013.10.013. Epub 2013 Oct 18. PMID 24145207
- [Result] Plaghki L, Mouraux A. How do we selectively activate skin nociceptors with a high power infrared laser? Physiology and biophysics of laser stimulation. Neurophysiol Clin. 2003 Dec;33(6):269-77. doi: 10.1016/j.neucli.2003.10.003. PMID 14678841
- [Result] Ravn P, Frederiksen R, Skovsen AP, Christrup LL, Werner MU. Prediction of pain sensitivity in healthy volunteers. J Pain Res. 2012;5:313-26. doi: 10.2147/JPR.S33925. Epub 2012 Aug 29. PMID 23055774